CLINICAL TRIAL: NCT02966002
Title: Aspirin as a Novel Anti-Inflammatory Modality in the Fontan Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated due to inability to recruit sufficient patients.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Adam Lubert, Clinical Instructor, Pediatric Cardiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00100325
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Fontan Procedure
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Intervention: aspirin (Experimental): 650 mg. Twice a day for 8 weeks
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
Patients who have undergone the Fontan procedure (a congenital heart surgery) may develop complications many years after their operation. Studies have shown that some of these patients develop an ongoing inflammatory state, which may be the cause of these late complications. Aspirin is a common over the counter anti-inflammatory medication used for many other chronic diseases. This study may help determine if aspirin therapy can limit the inflammation seen in Fontan patients and prevent these late complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have Fontan repair of single ventricle

Exclusion Criteria: Persons with the following history, conditions, or behavior will be excluded

* Active protein losing enteropathy within the past three years
* Congestive heart failure
* Active arrhythmias
* Taking Coumadin (Warfarin)
* Bleeding disorder
* Known esophageal varicies
* Consuming more than 10 alcoholic drinks per week.
* Pregnant
* Planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lubert, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Aspirin: 650 mg. Twice a day for 8 weeks
  Aspirin
Period: Overall Study
Arm/Group | Intervention: Aspirin
Started | 9
Completed | 5
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention: Aspirin
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 138.6 (16.6)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 47.6 (15.1)
High Sensitivity C-Reactive Protein [Mean (Standard Deviation); unit: mg/dL] | 0.24 (0.10)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Short-Form 36-Item Health Survey (SF-36) is a standardized health survey consisting of 36 questions that measure 8 dimensions of general health-related quality of life: physical functioning, role limitation due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and general mental health. The score is represented as an average of the individual question scores, and ranges from 0 (not functioning) to 100 (highest functioning). Higher scores indicate a better health status.
  units on a scale | 82.4 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Cholesterol
Description: Change will be measured from baseline to retest after 8 weeks of treatment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention: Aspirin
Number analyzed (Participants) | 5
mg/dL | -0.6 (15.5)
Statistical Analysis 1: Comparison: Intervention: Aspirin; Test type: Other; p = 0.96, t-test, 2 sided

2. Primary Outcome: Change in HDL (High-Density Lipoprotein)-Cholesterol
Description: Change will be measured from baseline to retest after 8 weeks of treatment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention: Aspirin
Number analyzed (Participants) | 5
mg/dL | 0.4 (17.3)
Statistical Analysis 1: Comparison: Intervention: Aspirin; Test type: Other; p = 0.67, t-test, 2 sided

3. Secondary Outcome: High Sensitivity CRP(C-Reactive Protein)
Description: Change will be measured from baseline to retest after 8 weeks of treatment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention: Aspirin
Number analyzed (Participants) | 5
mg/dL | 0.06 (0.09)
Statistical Analysis 1: Comparison: Intervention: Aspirin; Test type: Other; p = 0.18, t-test, 2 sided

4. Secondary Outcome: Quality of Life
Description: The Medical Outcomes Short-Form 36-Item Health Survey (SF-36) is a standardized health survey consisting of 36 questions that measure 8 dimensions of general health-related quality of life: physical functioning, role limitation due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and general mental health. The score is represented as an average of the individual question scores, and ranges from 0 (not functioning) to 100 (highest functioning). Higher scores indicate a better health status.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention: Aspirin
Number analyzed (Participants) | 5
units on a scale | 86.5 (4.1)
Statistical Analysis 1: Comparison: Intervention: Aspirin; Test type: Other; p = 0.25, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention: Aspirin
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention: Aspirin (N=5)
Bloody Bowel Movement (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT02966002/Prot_SAP_000.pdf